CLINICAL TRIAL: NCT01051050
Title: Using Wikis to Improve the Dissemination, Evaluation, and Application of Evidence-Based Medicine in Surgical Practice
Brief Title: Use of Wikis and Evidence-Based Medicine in Surgical Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HSC-MS-09-0573
Record Dates: First submitted 2010-01-14; First posted 2010-01-18 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Evidence Based Medicine
Keywords: Evidence based medicine; Improving surgical residents skills and application of EBM in surgical practice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mandatory use of surgery wiki (Other): Mandatory participation in journal club wiki which will include adding to and reviewing the information posted on the wiki. Contribution to the wiki will be required at least once during the study period.
  Interventions: Behavioral: Mandatory use of surgery wiki
- Voluntary use of surgery wiki (Other): Voluntary participation in the journal club wiki
  Interventions: Behavioral: Voluntary use of the surgery wiki

INTERVENTIONS:
Behavioral: Mandatory use of surgery wiki — Mandatory participation in the surgery wiki. This will include adding to and reviewing information posted on the wiki. Contribution of an evidence-based review will be required at least once during the study period.
  Arms: Mandatory use of surgery wiki
Behavioral: Voluntary use of the surgery wiki — Voluntary participation in the surgery wiki. Participants can choose to use the information in the wiki as well as contribute to the wiki.
  Arms: Voluntary use of surgery wiki

SUMMARY:
The goal of this study is to improve surgical residents' skills in critically appraising the literature and to promote the dissemination and application of the best available evidence to surgical practice. The hypothesis is that mandatory participation, with faculty oversight, in a journal club wiki will improve the dissemination, evaluation, and application of evidence-based medicine (EBM) in a surgical residency program at University of Texas Health Science Center at Houston (UT-Houston).

DETAILED DESCRIPTION:
The translation of evidence-based medicine (EBM) to clinical practice requires training in literature searching and critical appraisal, which is particularly lacking in surgery. The demands of surgical residency coupled with the 80-hour work week make attendance at journal clubs suboptimal. Internet technology such as wikis, which are free user-friendly collaborative websites, may be a solution to improving resident participation in journal club-related activities, but their utility is highly dependent upon resident contributions and usage. We propose a pilot randomized trial of mandatory versus voluntary participation in a general surgery journal club wiki to verify its feasibility, sustainability, and impact on resident EBM skills as measured with a validated questionnaire. Secondary outcomes will include resident self-assessment of wiki usage and comfort with EBM skills and faculty-assessed resident application of these skills in weekly morbidity and mortality conferences. If the wiki is feasible and sustainable, then the project will be expanded to include other surgical disciplines and cohorts (i.e. students, fellows, other institutions, other medical disciplines) to ensure generalizability. If beneficial, wikis could not only improve resident EBM skills, but also have a halo effect on students and faculty, and ultimately wikis could improve patient care. The assembled multi-disciplinary and multi-institutional team has significant collective expertise in evidence-based medicine, medical education, library skills, and clinical trial design and analysis which are necessary for this project.

ELIGIBILITY:
Inclusion Criteria:

* General surgery residents at UT Health Science Center at Houston

Exclusion Criteria:

* Not a general surgery resident at UT Health Science Center at Houston

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in performance on a questionnaire | 1 year

SECONDARY OUTCOMES:
self-assessment of wiki usage | 1 year
use of EBM in daily practice before and after the trial | 1 year
comfort with critical appraisal of the literature using a 5-point Likert scale | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lillian S Kao, MD, MS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center-Houston, Houston, Texas, United States